CLINICAL TRIAL: NCT05250492
Title: Evaluation of Analgesia by PENG Block Versus Intra-Articular Infiltration in Prosthetic Hip Surgery
Brief Title: Evaluation of Analgesia by PENG Block Versus Intra-Articular Infiltration in Prosthetic Hip Surgery (API)
Acronym: API
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-A00539-32
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2022-02

CONDITIONS: Hip Prosthesis; Analgesia; PENG Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with PENG block (Experimental)
  Interventions: Procedure: Prosthetic hip surgery
- Patients with intra-articular infiltration (Active Comparator)
  Interventions: Procedure: Prosthetic hip surgery

INTERVENTIONS:
Procedure: Prosthetic hip surgery — Total hip prosthesis performed by an anterior approach with intra-articular infiltration of an anesthetic product intraoperatively.
  OR
  - Total hip prosthesis performed by an anterior approach with infiltration of the same anesthetic product by ultrasound-guided PENG block intraoperatively.

SUMMARY:
The main objective of this study is to compare the effectiveness of the ultrasound-guided PENG block technique compared to intra-articular infiltration on postoperative morphine consumption during hip prosthetic surgery via the anterior minimally invasive approach under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old.
* Patient scheduled for anterior hip prosthesis.
* Affiliated patient or beneficiary of a social security scheme.
* Patient having been informed and having signed a free and informed consent.

Exclusion Criteria:

* Patient with a contraindication to local anesthesia.
* Patient with a high level of dependence, defined by level 1 or 2 of the Iso-Ressources Group (GIR).
* Patient participating in another clinical study.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of freedom by judicial or administrative decision.
* Pregnant, breastfeeding or parturient woman.
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption in the postoperative care unit | 1 hour
  Postoperative morphine consumption (in mg) in the postoperative care unit

SECONDARY OUTCOMES:
Postoperative morphine équivalent consumption at postoperative day 1 | 1 day
  postoperative morphine équivalent consumption (in mg) at postoperative day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Jean-François Oudet, Lanester, France